CLINICAL TRIAL: NCT03688776
Title: CSD1805: A Single-blind, Two-way Crossover Study to Assess Nicotine Uptake and Product Use Behavior in Moist Snuff Consumers Using Two Moist Snuff Products
Brief Title: CSD1805: Study to Assess Nicotine Uptake and Product Use Behavior in Moist Snuff Consumers Using Two Moist Snuff Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Collaborators: ICON Clinical Research Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CSD1805
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1805AA, 1805AB Use Group (Experimental): Use of product 1805AA exclusively for approximately 3 days prior to a PK assessment, followed by use of product 1805AB exclusively for approximately 3 days prior to a PK assessment.
  Interventions: Other: 1805AA; Other: 1805AB
- 1805AB, 1805AA Use Group (Experimental): Use of product 1805AB exclusively for approximately 3 days prior to a PK assessment, followed by use of product 1805AA exclusively for approximately 3 days prior to a PK assessment.
  Interventions: Other: 1805AA; Other: 1805AB

INTERVENTIONS:
Other: 1805AA — A moist snuff product
Other: 1805AB — A moist snuff product

SUMMARY:
The purpose of this study is to compare nicotine uptake and product use behavior during and following use of two moist snuff products in generally healthy, adult moist snuff users.

DETAILED DESCRIPTION:
This will be an single-blind, multi-center, randomized, two-way crossover study, conducted in generally healthy, adult moist snuff users who will be randomly assigned to the order in which they will use two moist snuff study products (comparator product, test product). The study will evaluate pharmacokinetic (PK) measures for two moist snuff products in a 7-day confinement setting.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English;
* Generally healthy male or female, 21 to 60 years of age, inclusive, at the time of signing informed consent;
* Positive urine cotinine test at the Screening Visit and Day 1;
* Females must be willing to use a form of contraception acceptable to the Principal Investigator (PI) from the time of signing the ICF until study discharge;
* Subjects' primary tobacco product must be a moist snuff product. Dual use of other forms of tobacco- and/or nicotine-containing products will be allowed but not more frequently than four days per week;
* Self-reports currently using at least one can of their non-pouched usual brand (UB) moist snuff per week for at least 3 months prior to Enrollment;
* Agrees to exclusively use the IP and not use any other tobacco- or nicotine-containing product during the course of the study;
* Able to safely perform the required study procedures, as determined by the PI.

Exclusion Criteria:

* Presence of clinically significant or unstable/uncontrolled acute or chronic medical conditions at the time of signing the ICF, as determined by the PI, that would preclude a subject from participating safely in the study (e.g., uncontrolled hypertension, cardiac disease, neurological disease, psychiatric disorders) based on safety assessments such as clinical laboratory tests, pregnancy tests, medical history, and physical/oral examinations;
* History, presence of, or clinical laboratory test results indicating diabetes;
* Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95mmHg, measured after being seated for 5 minutes;
* Hemoglobin level < 12.5 g/dL for females and < 13.0 g/dL for males at the Screening Visit;
* Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV);
* Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed;
* Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within 30 days prior to signing the ICF;
* History or presence of bleeding or clotting disorders;
* Any use of anticoagulants or aspirin (>325mg/day);
* Whole blood donation within 8 weeks (≤ 56 days) prior to the signing the ICF;
* Plasma donation within (≤) 7 days of signing the ICF;
* Participation in another clinical trial within (≤) 30 days of signing the ICF (the 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study);
* Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study;
* Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy;
* A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at the Screening Visit or Day 1;
* Postponing a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or a previous quit attempt within (≤) 30 days prior to signing the ICF;
* Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol test result at the Screening Visit or Day 1;
* Employed by a tobacco- or other nicotine-product manufacturing company, or the study site;
* Determined by the PI to be inappropriate for the study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
AUCnic 0-240 | -5, -1, 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90, 120, 150, 180, 210 and 240 Minutes
  area under the baseline-adjusted nicotine concentration- versus-time curve from time zero to 240 minutes after the start of Investigational Product (IP) use

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel DeNoia, MD, Principal Investigator — ICON Clinical Research; Melanie Fein, MD, Principal Investigator — High Point Clinical Trial Center
Locations (2):
- United States (2):
  - High Point Clinical Trials Center, High Point, North Carolina
  - ICON Clinical Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No